CLINICAL TRIAL: NCT01576341
Title: Open Label, Single Arm, Multicenter Study to Evaluate the Safety and Immunogenicity of HX575 Epoetin Alfa in the Treatment of Anemia Associated With Chronic Kidney Disease in Pre-dialysis and Dialysis Patients
Brief Title: HX575 Epoetin Alfa Subcutaneously (s.c.) in Chronic Kidney Disease (CKD)
Acronym: SENSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX575-308; 2011-002871-40 (EudraCT Number)
Record Dates: First submitted 2012-04-05; First posted 2012-04-12 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-04

CONDITIONS: Chronic Kidney Disease
Keywords: Epoetin alfa, ESA, HX575, CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HX575 epoetin alfa (Sandoz) (Experimental): Single arm
  Interventions: Drug: HX575 epoetin alfa (Sandoz)

INTERVENTIONS:
Drug: HX575 epoetin alfa (Sandoz) — Eligible patients are scheduled to receive HX575 (INN: Epoetin alfa) as a solution for injection in order to achieve or maintain the correction of renal anemia.
  Other Names: Binocrit®, Epoetin alfa HEXAL®, Novicrit®, Abseamed®

SUMMARY:
The study will assess the immunogenicity, safety, and efficacy of HX575 epoetin alfa administered subcutaneously (s.c.) in patients suffering from anemia due to chronic kidney disease (CKD)

ELIGIBILITY:
Main Inclusion Criteria:

* Adult male and female patients w or w/o dialysis treatment
* Stable i.v. or s.c. maintenance therapy with an EU-approved ESA treatment or ESA naïve.
* Adequate iron substitution

Main Exclusion Criteria:

* History of Pure Red Cell Aplasia (PRCA) or anti-erythropoietin (EPO) antibodies
* Contraindications for ESA therapy
* Serum albumin < 3.0 g/dL
* Immunocompromized patients (immunosuppressive treatment, chemotherapy)
* Hepatitis C infection on an active treatment or hepatitis B or human immunodeficiency virus (HIV) infection
* Systemic lupus erythematosus
* Symptomatic congestive heart failure, Unstable angina pectoris, or myocardial infarction within 6 months
* History of malignancy of any organ system within the last 5 years
* History of use of any non-EU approved ESA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2012-04; Primary Completion 2014-10 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceuticals, Study Chair — Sandoz
Locations (50):
- Germany (3):
  - Sandoz Investigative Site, Düsseldorf
  - Sandoz Investigative Site, Homberg (Efze)
  - Sandoz Investigative Site, Nettetal
- Sandoz Investigative Site, Bari, Italy
- Poland (8):
  - Sandoz Investigative Site, Częstochowa
  - Sandoz Investigative Site, Gdansk
  - Sandoz Investigative Site, Gdynia
  - Sandoz Investigative Site, Olkusz
  - Sandoz Investigative Site, Poznan
  - Sandoz Investigative Site, Płock
  - Sandoz Investigative Site, Wadowice
  - Sandoz Investigative Site, Warzawa
- Romania (5):
  - Sandoz Investigative Site, Bucharest
  - Sandoz Investigative Site, Constanța
  - Sandoz Investigative Site, Lasi
  - Sandoz Investigative Site, Oradea
  - Sandoz Investigative Site, Timișoara
- Russia (17):
  - Sandoz Investigative Site, Chelyabinsk
  - Sandoz Investigative Site, Kemerovo
  - Sandoz Investigative Site, Kolomna
  - Sandoz Investigative Site, Moscow
  - Sandoz Investigative Site, Mytischi
  - Sandoz Investigative Site, Nizhny Novgorod
  - Sandoz Investigative Site, Novosibirsk
  - Sandoz Investigative Site, Orenburg
  - Sandoz Investigative Site, Petrozavodsk
  - Sandoz Investigative Site, Podolsk
  - Sandoz Investigative Site, Pyatigorsk
  - Sandoz Investigative Site, Ryazan
  - Sandoz Investigative Site, Saint Petersburg
  - Sandoz Investigative Site, Saratov
  - Sandoz Investigative Site, Smolensk
  - Sandoz Investigative Site, Yaroslavl
  - Sandoz Investigative Site, Yekaterinburg
- Turkey (Türkiye) (3):
  - Sandoz Investigative Site, Adana
  - Sandoz Investigative Site, Ankara
  - Sandoz Investigative Site, Istanbul
- Ukraine (13):
  - Sandoz Investigative Site, Chernivtsi
  - Sandoz Investigative Site, Dnipropetrovsk
  - Sandoz Investigative Site, Donetsk
  - Sandoz Investigative Site, Ivano-Frankivsk
  - Sandoz Investigative Site, Kharkiv
  - Sandoz Investigative Site, Kyiv
  - Sandoz Investigative Site, Luhansk
  - Sandoz Investigative Site, Mykolayiv
  - Sandoz Investigative Site, Poltava
  - Sandoz Investigative Site, Ternopil
  - Sandoz Investigative Site, Uzhhorod
  - Sandoz Investigative Site, Zaporizhya
  - Sandoz Investigative Site, Zhitomyr

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients, suffering from anemia associated with chronic Kidney Disease (CKD), were treated s.c. with HX575 at least once per week in order to achieve and maintain Hb concentration within the target range of 10.0 to 12.0 g/dL. 417 patients were enrolled.
Pre-assignment Details: Male and female patients (ESA [Erythropoiesis Stimulating Agent]-naïve/on ESA-maintenance therapy, i.v./s.c.) aged 18 years/older, suffering from anemia assoc. with CKD, with/without dialysis treatment. Anemia: Mean Hb conc. <= 11.0 g/dL for ESA naïve, 9.0-12.0 g/dL for patients receiving ESA therapy.
Groups:
- HX575, Safety Population: In the single arm study, HX575 was tested as investigational medicinal product. The single arm includes ESA-naïve patients and patients on ESA-maintenance therapy.
Period: Overall Study
Arm/Group | HX575, Safety Population
Started | 417
Completed | 324
Not Completed | 93
Not completed — Withdrawal by Subject | 24
Not completed — Adverse Event | 10
Not completed — Death | 21
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 2
Not completed — Kidney transplantation | 10
Not completed — Protocol Violation | 12
Not completed — Other | 12

BASELINE CHARACTERISTICS:
Population: Safety population: The safety population consists of all patients that received at least one dose of study drug
Groups:
- HX575, Safety Population: The Study was designed as single arm study with HX575 tested as investigational medicinal product. The safety population (SAF) consisted of all patients that received at least one dose of study drug. 417 patients enrolled, 416 treated. Group includes ESA-naïve patients and patients on ESA-maintenance therapy.
Arm/Group | HX575, Safety Population
Number analyzed (Participants) | 416
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (15.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 198
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 416
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russian Federation | 107
  Romania | 40
  Turkey | 33
  Ukraine | 179
  Poland | 47
  Italy | 5
  Germany | 5
Height [Mean (Standard Deviation); unit: cm] | 166.9 (9.44)
Weight [Mean (Standard Deviation); unit: kg] | 70.6 (15.92)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.26 (5.073)
ESA pre-treatment [Number; unit: participants] — A patient is considered to be ESA naïve if the patient did not receive any ESA therapy within 2 months prior to first screening visit.
  participants
    ESA naive | 250
    ESA maintenance | 166

OUTCOME MEASURES:

1. Primary Outcome: Anti-Erythropoietin (EPO) Antibodies
Description: The incidence of antibody formation against epoetin in Radio-immuno-precipitation (RIP) assay
Time Frame: 52 weeks
Population: Safety population: The safety population consists of all patients that received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HX575: HX575 administered s.c. at least once per week. During the treatment period the dose was individually titrated to maintain hemoglobin levels between 10.0 and 12.0 g/dL
Arm/Group | HX575
Number analyzed (Participants) | 416
percentage of participants | 1.7 [0.7 to 3.4]
Statistical Analysis 1: Comparison: HX575; Test type: Other; Incidence rate = 0.019 — Incidence rate is based on duration of treatment period (years)

2. Secondary Outcome: Hemoglobin Level and Change From Baseline Period at Visit 16 (End of Study)
Description: Actual values of hemoglobin levels at end of study visit and change from Baseline Period (Week -4 to Week -1)
Time Frame: 52 weeks
Population: Per-protocol population (all patients that received at least one dose of study drug) with non-missing Hemoglobin value at Visit 16 (end of study).
Measure: Mean (Standard Deviation); unit: g/dL
Groups:
- HX575 - ESA Naive: HX575 administered s.c. at least once per week. During the treatment period the dose was individually titrated to maintain hemoglobin levels between 10.0 and 12.0 g/dL. At study start patients were either ESA (Erythropoiesis Stimulating Agent) naive or on ESA maintenance treatment. This group only contains patients that were ESA naive at study start, e.g. did not receive any ESA dose within 2 months prior to first screening visit.
- HX575 - ESA Maintenance: HX575 administered s.c. at least once per week. During the treatment period the dose was individually titrated to maintain hemoglobin levels between 10.0 and 12.0 g/dL. At study start patients were either ESA (Erythropoiesis Stimulating Agent) naive or on ESA maintenance treatment. This group only contains patients that were on ESA maintenance treatment at study start, e.g. did receive at least one dose of commercial ESA treatment within 2 months prior to first screening visit.
Arm/Group | HX575 - ESA Naive | HX575 - ESA Maintenance | HX575
Number analyzed (Participants) | 199 | 144 | 343
g/dL
  Actual Value | 10.81 (1.336) | 10.86 (1.060) | 10.83 (1.226)
  Change from Baseline Period | 1.61 (1.601) | 0.22 (1.223) | 1.02 (1.606)

ADVERSE EVENTS:
Time Frame: 4 weeks (screening period) + 52 weeks (treatment period)
Groups:
- HX575, Safety Population: Study was designed as single arm study with HX575 tested as investigational medicinal product. Safety population includes ESA therapy naïve patients and ESA maintenance patients. Shown are all AEs including non-treatment related AEs.
Arm/Group | HX575, Safety Population
All-Cause Mortality (participants affected / at risk) | 25/416
Serious Adverse Events (participants affected / at risk) | 103/416
Other Adverse Events (participants affected / at risk) | 121/416
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575, Safety Population (N=416)
Anaemia (Blood and lymphatic system disorders) | 1 (1) — † A
Acute coronary syndrome (Cardiac disorders) | 2 (2) — † A
Acute left ventricular failure (Cardiac disorders) | 1 (1) — † A
Acute myocardial infarction (Cardiac disorders) | 2 (2) — † A
Angina pectoris (Cardiac disorders) | 3 (3) — † A
Angina unstable (Cardiac disorders) | 2 (3) — † A
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) — † A
Atrial fibrillation (Cardiac disorders) | 2 (2) — † A
Atrial tachycardia (Cardiac disorders) | 1 (1) — † A
Cardiac arrest (Cardiac disorders) | 1 (1) — † A
Cardiac failure (Cardiac disorders) | 2 (2) — † A
Cardiac failure acute (Cardiac disorders) | 1 (1) — † A
Cardiac failure chronic (Cardiac disorders) | 1 (1) — † A
Cardiomyopathy (Cardiac disorders) | 1 (1) — † A
Cardiovascular insufficiency (Cardiac disorders) | 2 (2) — † A
Carditis (Cardiac disorders) | 1 (1) — † A
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) — † A
Coronary artery stenosis (Cardiac disorders) | 1 (1) — † A
Myocardial infarction (Cardiac disorders) | 5 (5) — † A
Myocardial ischaemia (Cardiac disorders) | 1 (1) — † A
Myocarditis (Cardiac disorders) | 1 (1) — † A
Adrenal mass (Endocrine disorders) | 1 (1) — † A
Hyperparathyroidism (Endocrine disorders) | 1 (1) — † A
Hyperparathyroidism secondary (Endocrine disorders) | 2 (2) — † A
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) — † A
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) — † A
Gastritis (Gastrointestinal disorders) | 1 (1) — † A
Gastritis erosive (Gastrointestinal disorders) | 1 (2) — † A
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 (1) — † A
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) — † A
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) — † A
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1) — † A
Oesophagitis (Gastrointestinal disorders) | 1 (1) — † A
Pancreatitis (Gastrointestinal disorders) | 1 (1) — † A
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) — † A
Calcinosis (General disorders) | 1 (1) — † A
Death (General disorders) | 1 (1) — † A
Multi-organ failure (General disorders) | 1 (1) — † A
Systemic inflammatory response syndrome (General disorders) | 1 (1) — † A
Bile duct stone (Hepatobiliary disorders) | 1 (1) — † A
Hypersensitivity (Immune system disorders) | 1 (1) — † A
Acute hepatitis b (Infections and infestations) | 1 (1) — † A
Appendicitis (Infections and infestations) | 1 (1) — † A
Bronchopneumonia (Infections and infestations) | 2 (2) — † A
Carbuncle (Infections and infestations) | 1 (1) — † A
Cellulitis (Infections and infestations) | 1 (1) — † A
Device related infection (Infections and infestations) | 2 (3) — † A
Endocarditis (Infections and infestations) | 1 (1) — † A
Erysipelas (Infections and infestations) | 1 (1) — † A
Intervertebral discitis (Infections and infestations) | 2 (2) — † A
Laryngitis (Infections and infestations) | 1 (1) — † A
Lobar pneumonia (Infections and infestations) | 1 (1) — † A
Orchitis (Infections and infestations) | 1 (1) — † A
Osteomyelitis (Infections and infestations) | 1 (1) — † A
Peritonitis (Infections and infestations) | 5 (6) — † A
Pneumonia (Infections and infestations) | 5 (5) — † A
Pyelonephritis chronic (Infections and infestations) | 1 (1) — † A
Sepsis (Infections and infestations) | 1 (1) — † A
Staphylococcal sepsis (Infections and infestations) | 1 (1) — † A
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) — † A
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) — † A
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) — † A
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) — † A
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) — † A
Shunt occlusion (Injury, poisoning and procedural complications) | 1 (1) — † A
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) — † A
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) — † A
Acidosis (Metabolism and nutrition disorders) | 1 (1) — † A
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) — † A
Dehydration (Metabolism and nutrition disorders) | 1 (1) — † A
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) — † A
Fluid retention (Metabolism and nutrition disorders) | 1 (1) — † A
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) — † A
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) — † A
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — † A
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1) — † A
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — † A
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — † A
Cerebral haemorrhage (Nervous system disorders) | 1 (1) — † A
Cerebrovascular accident (Nervous system disorders) | 3 (3) — † A
Extrapyramidal disorder (Nervous system disorders) | 1 (1) — † A
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) — † A
Ischaemic stroke (Nervous system disorders) | 1 (1) — † A
Transient ischaemic attack (Nervous system disorders) | 1 (1) — † A
Uraemic encephalopathy (Nervous system disorders) | 1 (1) — † A
Azotaemia (Renal and urinary disorders) | 2 (2) — † A
Diabetic nephropathy (Renal and urinary disorders) | 1 (2) — † A
Renal cyst (Renal and urinary disorders) | 1 (1) — † A
Renal failure (Renal and urinary disorders) | 2 (2) — † A
Renal failure chronic (Renal and urinary disorders) | 20 (24) — † A
Urinary retention (Renal and urinary disorders) | 1 (1) — † A
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (2) — † A
Metrorrhagia (Reproductive system and breast disorders) | 2 (2) — † A
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) — † A
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 (2) — † A
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — † A
Arteriosclerosis (Vascular disorders) | 1 (2) — † A
Extremity necrosis (Vascular disorders) | 1 (1) — † A
Haematoma (Vascular disorders) | 1 (1) — † A
Hypertension (Vascular disorders) | 5 (5) — † A
Hypertensive crisis (Vascular disorders) | 2 (2) — † A
Hypertensive emergency (Vascular disorders) | 1 (1) — † A
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HX575, Safety Population (N=416)
Diarrhoea (Gastrointestinal disorders) | 9 (11) — † A
Oedema peripheral (General disorders) | 9 (13) — † A
Nasopharyngitis (Infections and infestations) | 13 (15) — † A
Pneumonia (Infections and infestations) | 10 (13) — † A
Urinary tract infection (Infections and infestations) | 9 (11) — † A
Hyperkalaemia (Metabolism and nutrition disorders) | 19 (25) — † A
Renal failure chronic (Renal and urinary disorders) | 39 (42) — † A
Hypertension (Vascular disorders) | 42 (75) — † A

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.